CLINICAL TRIAL: NCT05354141
Title: Bone Marrow Mesenchymal Stem Cell Derived Extracellular Vesicles for Hospitalized Patients With Moderate-to-Severe ARDS: A Phase III Clinical Trial
Brief Title: Extracellular Vesicle Treatment for Acute Respiratory Distress Syndrome (ARDS) (EXTINGUISH ARDS)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Direct Biologics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DB-EF-PHASEIII-0001
Record Dates: First submitted 2022-04-27; First posted 2022-04-29 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Acute Respiratory Distress Syndrome; ARDS
Keywords: ExoFlo; Extracellular Vesicles; Exosome; ARDS
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized, double-blinded, placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-Blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Normal saline 100 mL
  Interventions: Other: Intravenous normal saline
- Experimental Dose (Experimental): Normal saline 85 mL and ExoFlo 15 mL
  Interventions: Biological: ExoFlo

INTERVENTIONS:
Biological: ExoFlo — Intravenous administration of bone marrow mesenchymal stem cell derived extracellular vesicles
  Arms: Experimental Dose
Other: Intravenous normal saline — Placebo
  Arms: Placebo

SUMMARY:
To evaluate the safety and efficacy of intravenous (IV) administration of bone marrow mesenchymal stem cell derived extracellular vesicles (EVs), ExoFlo, versus placebo for the treatment of hospitalized patients with moderate-to-severe Acute Respiratory Distress Syndrome (ARDS).

DETAILED DESCRIPTION:
This is a Phase III, multicenter, randomized, double-blinded, placebo-controlled trial for the treatment of moderate-to-severe Acute Respiratory Distress Syndrome (ARDS).

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18-75 years of age
2. Presence of the following criteria for moderate to severe ARDS as defined by the Berlin Criteria within 24 hours of the first infustion:

   1. Onset within 7 days of known clinical insult or requiring increasing respiratory rate, increasing oxygen flows, or increased work of breathing, and
   2. Bilateral lung opacities not fully explained by pleural effusions, atelectasis, or nodules, and
   3. PaO2/FiO2 (P/F ratio) ≤ 200 mm Hg, and
   4. Invasive or noninvasive ventilation with a minimum PEEP 5 cm H2O or minimum of continuous positive airway pressure (CPAP) 5 cm H2O, or High Flow Nasal Oxygen at ≥ 30 L/min, and
   5. Respiratory failure not fully explained by cardiac failure or fluid overload.

Exclusion Criteria:

1. Lack of signed and dated informed consent form (either by the individual or by the individual's healthcare proxy).
2. Stated unwillingness to comply with all study procedures and availability for the duration of the study
3. Vulnerable populations such as pregnant patients, children, individuals with severe physical or mental disabilities who cannot provide meaningful consent.
4. Active malignancy requiring treatment within the last two years, with the exception of non-melanoma skin cancers.
5. Major physical trauma in the last 2 days, including motor vehicle accidents, assaults, mechanical falls with sequelae of significant bleeding or craniofacial bruising, and surgeries, such that not one or more injury may be undiagnosed at time of screening.
6. Duration of mechanical ventilation exceeds 3 days or 72 hours from diagnosis of ARDS.
7. ALT or AST > 8 x Upper Limit of Normal (ULN).
8. Documented history of cirrhosis.
9. DNR order, as in electing not to receive chest compressions, cardiac defibrillation, cardiac drugs, or intubation.
10. Moribund-expected survival < 24 hours.
11. Severe metabolic disturbances at randomization (e.g., ketoacidosis, pH < 7.2)
12. Patient currently connected to Extracorporeal Membrane Oxygenation at initiation of screening.
13. If the candidate, either a male or female of reproductive potential, is unwilling to two methods of highly effective birth control contraception such as condoms with oral contraceptive pill or choose to remain abstinent if already practicing abstinence during the screening period. The required duration of usage of double method OR maintenance of abstinence must include the time from the beginning of the screening period until Day 61, day of withdrawal or early termination
14. Use of investigational COVID-19 agents or any other investigational agents within 30 days prior to the first dose.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 970 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of 60-day All-cause Mortality | 60 days
  To evaluate the 60-day mortality rate for IMP 15mL as a treatment for moderate-to-severe ARDS compared to placebo. Reducing the mortality rate for hospitalized patients with moderate-to-severe ARDS is a measure of the treatment effect.

SECONDARY OUTCOMES:
Time to death | 60 days
  Reducing the mortality rate for hospitalized patients moderate-to-severe ARDS is a measure of the treatment effect.
Ventilator-free days (VFDs) | Day 29
  Number of days for which patients are not on mechanical ventilation.
Oxygen free days | Day 29
  Number of days for which patients are not on oxygen support.
ICU free days | Day 29
  Number of days for which patients are not in the ICU.
Incidence of Treatment Emergent Serious Adverse Events (TESAEs) | 61 days
  Safety comparison performed between IMP 15 mL and placebo arms

CONTACTS AND LOCATIONS:
Overall Officials: Bill Arana, Study Director — Direct Biologics, LLC
Locations (38):
- United States (38):
  - Direct Biologics Investigational Site, Birmingham, Alabama
  - Direct Biologics Investigational Site, Chandler, Arizona
  - Direct Biologics Investigational Site, Phoenix, Arizona
  - Direct Biologics Investigational Site, Little Rock, Arkansas
  - Direct Biologics Investigational Site, Davis, California
  - Direct Biologics Investigational Site, Fullerton, California
  - Direct Biologics Investigational Site, Irvine, California
  - Direct Biologics Investigational Site, Orange, California
  - Direct Biologics Investigational Site, Sacramento, California
  - Direct Biologics Investigational Site, San Francisco, California
  - Direct Biologics Investigational Site, Washington D.C., District of Columbia
  - Direct Biologics Investigational Site, Jacksonville, Florida
  - Direct Biologics Investigational Site, Boise, Idaho
  - Direct Biologics Investigational Site, Iowa City, Iowa
  - Direct Biologics Investigational Site, Wichita, Kansas
  - Direct Biologics Investigational Site, Silver Spring, Maryland
  - Direct Biologics Investigational Site, Boston, Massachusetts
  - Direct Biologics Investigational Site, Burlington, Massachusetts
  - Direct Biologics Investigational Site, Springfield, Massachusetts
  - Direct Biologics Investigational Site, Ann Arbor, Michigan
  - Direct Biologics Investigational Site, Detroit, Michigan
  - Direct Biologics Investigational Site, Jackson, Mississippi
  - Direct Biologics Investigational Site, Flushing, New York
  - Direct Biologics Investigational Site, Queens, New York
  - Direct Biologics Investigational Site, The Bronx, New York
  - Direct Biologics Investigational Site, Durham, North Carolina
  - Direct Biologics Investigational Site, Winston-Salem, North Carolina
  - Direct Biologics Investigational Site, Cincinnati, Ohio
  - Direct Biologics Investigational Site, Cleveland, Ohio
  - Direct Biologics Investigational Site, Portland, Oregon
  - Direct Biologics Investigational Site, Charleston, South Carolina
  - Direct Biologics Investigational Site, Knoxville, Tennessee
  - Direct Biologics Investigational Site, Nashville, Tennessee
  - Direct Biologics Investigational Site, Dallas, Texas
  - Direct Biologics Investigational Site, Fort Worth, Texas
  - Direct Biologics Investigational Site, Houston, Texas
  - Direct Biologics Investigational Site, Murray, Utah
  - Direct Biologics Investigational Site, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Direct Biologics, LLC — https://directbiologics.com/